CLINICAL TRIAL: NCT06889753
Title: A Randomized, Triple-blind, Placebo Controlled, Parallel Clinical Trial to Investigate the Effect of Pollen Extracts on Menopausal Symptoms in Healthy Women.
Brief Title: A Clinical Trial to Investigate the Effect of Pollen Extracts on Menopausal Symptoms in Healthy Women.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Graminex LLC (Other)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24GXCFG01
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-03

CONDITIONS: Menopausal Women
Keywords: Menopause; Flower Pollen Extracts; Water Soluble Pollen Extract; Lipid Soluble Pollen Extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Graminex Water Soluble Pollen Extract (WSPE) (Experimental): Graminex WSPE is a water soluble extract from flower pollen standardized to 6% amino acids.
  Interventions: Dietary Supplement: Graminex WSPE
- Graminex Lipid Soluble Pollen Extract (LSPE) (Experimental): Graminex LSPE is a lipid soluble pollen extract standardized to 7% phytosterols.
  Interventions: Dietary Supplement: Graminex LSPE
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Graminex WSPE — Graminex Water Soluble Pollen Extract is standardized to 6% amino acids.
  Arms: Graminex Water Soluble Pollen Extract (WSPE)
Dietary Supplement: Graminex LSPE — Graminex Lipid Soluble Pollen Extract is standardized to 7% phytosterols.
  Arms: Graminex Lipid Soluble Pollen Extract (LSPE)
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this study is to investigate the effect of pollen extracts on menopausal symptoms in healthy women The main question it aims to answer is:

What is the difference in change in severity of menopausal symptoms as assessed by the total Menopause Rating Scale (MRS) score from baseline at Week 36 between Graminex Water Soluble Pollen Extract (WSPE), Lipid Soluble Pollen Extract (LSPE), and Placebo?

Participants will be asked to complete the MRS assessment tool to rate their menopausal symptoms while receiving either WSPE, LSPE, or Placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Females between 45-60 years of age, inclusive
2. BMI 18.5 kg/m2 - 34.9 kg/m2 inclusive
3. Self-reported menopausal women who have not had a menstrual period for >12 months prior to screening and are experiencing at least moderate menopausal symptoms as assessed by the total MRS score of ≥9 at screening
4. Presence of menopausal symptoms for at least six months prior to screening including, vasomotor symptoms (hot flushes, sweating) AND at least two of the following symptoms: sleep disturbance, joint pain, mood changes, fatigue and lack of energy, vaginal dryness, urinary changes, and changes in sexual function
5. Agrees to maintain current lifestyle as much as possible throughout the study, including diet, exercise, medications, dietary supplements, and sleep
6. Able and willing to complete all study assessments
7. Provided voluntary, written, informed consent to participate in the study
8. Healthy as determined by medical history with no unstable, diagnosed medical conditions as assessed by the Qualified Investigator (QI)

Exclusion Criteria:

1. Females who have had unilateral oophorectomy or hysterectomy or uterine ablation
2. Allergy (including bee products or pollen, sensitivity, or intolerance to investigational products or placebo ingredients
3. Ongoing diagnosis with anxiety disorder, sleep disorder, or major depression as assessed by the QI
4. Ongoing unstable diagnosis of musculoskeletal disorders as assessed by the QI
5. Current untreated urogenital diagnosis as assessed by the QI
6. Unstable metabolic disease or chronic diseases as assessed by the QI
7. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
8. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
9. Current unstable Type I or Type II diabetes
10. Significant cardiovascular event in the past six months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
11. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
12. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least three months will be considered by the QI
13. Major surgery in the past three months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
14. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years
15. after diagnosis are acceptable
16. Individuals with unstable autoimmune disease or are immune compromised as assessed by the QI
17. Use of medical cannabinoid products
18. Chronic use of cannabinoid products (>2 times/week) as assessed by the QI
19. Alcohol intake average of >2 standard drinks per day as assessed by the QI
20. Alcohol or drug abuse within the last 12 months
21. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy of the investigational product (Sections 7.3.1 and 7.3.2)
22. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
23. Individuals who are unable to give informed consent
24. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant
25. Asthmatic, as assessed by the QI

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The difference in change in severity of menopausal symptomsbaseline at Week 36 between Graminex WSPE, Graminex LSPE, and Placebo | Week 0 (baseline) to 36
  The difference in change in severity of menopausal symptoms as assessed by the total Menopause Rating Scale (MRS) score from baseline at Week 36 between Graminex WSPE, Graminex LSPE, and Placebo.

SECONDARY OUTCOMES:
The difference in change in severity of menopausal symptoms from baseline at Week 6 between Graminex WSPE, Graminex LSPE, and Placebo | Week 0 (baseline) to 6
  The difference in change in severity of menopausal symptoms as assessed by total MRS score from baseline at Week 6 between Graminex WSPE, Graminex LSPE, and Placebo.
The difference in change in severity of menopausal symptoms from baseline at Week 12 between Graminex WSPE, Graminex LSPE, and Placebo | Week 0 (baseline) to 12
  The difference in change in severity of menopausal symptoms as assessed by total MRS score from baseline at Week 12 between Graminex WSPE, Graminex LSPE, and Placebo.
The difference in change in severity of menopausal symptoms from baseline at Week 24 between Graminex WSPE, Graminex LSPE, and Placebo | Week 0 (baseline) to 24
  The difference in change in severity of menopausal symptoms as assessed by total MRS score from baseline at Week 24 between Graminex WSPE, Graminex LSPE, and Placebo.
The difference in change in scores of individual domains of the MRS including Somatic, Psychological, and Urogenital domains between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 6 | Week 0 (baseline) to 6
  The difference in change in scores of individual domains of the MRS including Somatic, Psychological, and Urogenital domains between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 6.
The difference in change in scores of individual domains of the MRS including Somatic, Psychological, and Urogenital domains between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 12 | Week 0 (baseline) to 12
  The difference in change in scores of individual domains of the MRS including Somatic, Psychological, and Urogenital domains between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 12.
The difference in change in scores of individual domains of the MRS including Somatic, Psychological, and Urogenital domains between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 24 | Week 0 (baseline) to 24
  The difference in change in scores of individual domains of the MRS including Somatic, Psychological, and Urogenital domains between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 24.
The difference in change in scores of individual domains of the MRS including Somatic, Psychological, and Urogenital domains between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 36 | Week 0 (baseline) to 36
  The difference in change in scores of individual domains of the MRS including Somatic, Psychological, and Urogenital domains between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 36.
The difference in change in scores of individual symptoms included in the MRS between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 6 | Week 0 (baseline) to 6
  The difference in change in scores of individual symptoms included in the MRS between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 6.
The difference in change in scores of individual symptoms included in the MRS between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 12 | Week 0 (baseline) to 12
  The difference in change in scores of individual symptoms included in the MRS between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 12.
The difference in change in scores of individual symptoms included in the MRS between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 24. | Week 0 (baseline) to 24
  The difference in change in scores of individual symptoms included in the MRS between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 24.
The difference in change in scores of individual symptoms included in the MRS between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 36 | Week 0 (baseline) to 36
  The difference in change in scores of individual symptoms included in the MRS between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 36
The difference in change in sleep disturbance between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 6 | Week 0 (baseline) to 6
  The difference in change in sleep disturbance as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance form 8b between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 6
The difference in change in sleep disturbance between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 12 | Week 0 (baseline) to 12
  The difference in change in sleep disturbance as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance form 8b between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 12.
The difference in change in sleep disturbance between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 24 | Week 0 (baseline) to 24
  The difference in change in sleep disturbance as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance form 8b between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 24.
The difference in change in sleep disturbance between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 36 | Week 0 (baseline) to 36
  The difference in change in sleep disturbance as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance form 8b between Graminex WSPE, Graminex LSPE, and Placebo from baseline at Week 36.

OTHER OUTCOMES:
Incidence of post-emergent adverse events (AE) | Week 0 (baseline) to 36
  Incidence of post-emergent adverse events (AE)
Clinically relevant changes in blood pressure (BP) after supplementation | Week 0 (baseline) to 36
  Clinically relevant changes in blood pressure (BP) after supplementation with WPSE
Clinically relevant changes in blood pressure (BP) after supplementation | Week 0 (baseline) to 36
  Clinically relevant changes in blood pressure (BP) after supplementation with LPSE
Clinically relevant changes in heart rate (HR) after supplementation | Week 0 (baseline) to 36
  Clinically relevant changes in heart rate (HR) after supplementation with WSPE
Clinically relevant changes in heart rate (HR) after supplementation | Week 0 (baseline) to 36
  Clinically relevant changes in heart rate (HR) after supplementation with LSPE

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No